CLINICAL TRIAL: NCT05700188
Title: Explore the Diagnosis and Treatment Outcome of Alimentary Tract Cancer in National Cheng Kung University Hospital
Brief Title: Outcome of GI Cancer in NCKUH
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-108-113
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2013-01

CONDITIONS: Collection of Real-world Data in a Single Institute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffin-embedded (FFPE) tissue sample before or after treatment will be collected for next generation sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Resectable: Patients with resectable pancreatic cancer
- Borderline resectable: Patients with borderline resectable pancreatic cancer
- Locally advanced: Patients with locally advanced unresectable pancreatic cancer
- Metastatic: Patients with metastatic pancreatic cancer

SUMMARY:
Alimentary tract cancer patients treated at National Cheng Kung University Hospital during 2013/01/01 to 2020/12/31 were reviewed.

DETAILED DESCRIPTION:
We would like to explore the treatment strategy and clinical outcome of alimentary tract cancer in National Cheng Kung University Hospital. The result could help physician to further realize the real world practice of cancer treatment in Taiwan and might also help clinician to optimize the diagnosis and treatment strategy in alimentary tract cancer patients. Alimentary tract cancer patients treated at National Cheng Kung University Hospital during 2013/01/01 to 2020/12/31.

ELIGIBILITY:
Inclusion Criteria:

All patients with pancreatic cancer treated at National Cheng Kung University Hospital during 2013/01/01 to 2020/12/31

Exclusion Criteria:

No treatment or refuse treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pancreatic cancer treated at National Cheng Kung University Hospital during 2013/01/01 to 2020/12/31 were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 10 years
  Overall survival of patient received study treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 10 years
  Progression-free survival of patient received study treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - National Institute of Cancer Research, Tainan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Su YY, Chao YJ, Wang CJ, Liao TK, Su PJ, Huang CJ, Chiang NJ, Yu YT, Tsai HM, Chen LT, Shan YS. The experience of neoadjuvant chemotherapy versus upfront surgery in resectable pancreatic cancer: a cross sectional study. Int J Surg. 2023 Sep 1;109(9):2614-2623. doi: 10.1097/JS9.0000000000000495. PMID 37300888